## NCT03141281 Unique Protocol ID: 2017.20622 Date: 08/19/2019

## INFORMED CONSENT FORM (Participants for laboratory studies from the community)

I freely and voluntarily and without element of force or coercion, consent to be a participant in the research project entitled "Technology-Based Cognitive Interventions: Comparative Effectiveness and Adherence". This research is being conducted by Drs. Walter Boot and Neil Charness, who are researchers at the Florida State University.

I understand the purpose of their research project is to better understand how training programs are related to driving skill and/or cognition. As a participant in this study, you may be asked to complete questionnaires asking for demographic information such as age, gender, and work history, as well as questionnaires about Computer and Internet Experience and Attitudes towards Computers, and questionnaires about independence, well-being, knowledge of financial fraud and driving simulators, and quality of life. You may also be asked to complete simulated driving tasks such as making a left turn at an intersection, passing cyclists riding on the side of the road, and reacting to traffic signals using an electronic driving simulator located in the laboratory. Additionally, tests measuring perceptual, cognitive and psychomotor abilities may be administered. I understand that my involvement allows these researchers to recommend guidelines to minimize the risk to cognitive health, improve the safety of all drivers, and help reduce the risk of financial fraud.

As a participant in this study you may be asked to complete the questionnaires relating to technology, independence, well-being, social isolation, driving simulators, financial literacy, and quality of life for a second time approximately 1 month from today, and for a third time approximately 12 months from today. Additionally, you may be asked to complete the simulated driving tasks approximately 1 month from today and approximately 12 months from today. Other participants may only be asked to complete the study measures once without the need to return for follow-up measures.

As a participant in this study you may be assigned to have a laptop or an "All in One Touch Screen" tablet-based computer system to take home to complete additional training that may benefit your driving, cognitive, or financial skills. In this instance, you will be asked to complete a program on the tablet that may take up to 20 hours over the course of five weeks. The tablet device is to be returned after the training course is complete. Other participants may not be assigned a computer to take home or have any training course.

I understand that if I participate in the study, I will also receive information from the person who provided me with this form who will be able to describe which of the conditions above applies and will also provide details about the length of time the study will last. I understand my participation is totally voluntary and I may stop participation at any time. I understand that everything I say will be kept strictly confidential to the extent allowable by law. Any data that results from my participation will be made totally anonymous, and will not be attributable to any individual. I understand that I may be audio and video recorded by the researcher. Any recordings will be kept by the researcher on a password-protected computer. I understand that only the researcher

will have access to recordings if any are made and that the audio and video recordings will be destroyed five years after the study is complete.

I understand that there are seven features of the study process designed to maximize my confidentiality regarding audio and video recordings. These are described below.

- 1. I understand that I can review the data, including photographs, in order that any information I deem sensitive can be deleted from it. This decision is at my discretion.
- 2. I understand that I can withdraw from the study at any time, and have the data, including any video recordings, destroyed in my presence. This decision is at my discretion.
- 3. I understand that, at any time after the study, I can request that all data be destroyed in my presence obtained through my participation. This decision is at my discretion.
- 4. I understand that any video recordings that result from my participation will be marked only with an anonymous code and the name of the researcher that conducted the study.
- 5. I understand that any recording taken during my participation will be destroyed within five year of study completion.
- 6. All data, including any video recording, will be kept by the researcher in a locked filing cabinet and password-protected computer in the Psychology Department, Florida State University.
- 7. I understand that anonymous data will be stored in a searchable, electronic database that can be accessed by FSU and external researchers interested in reanalyzing the data. Any information in this data that could connect me will be deleted and replaced with a placeholder, such as 'person X'.

Participation in this study is voluntary and there are no significant risks to you. Any stress or discomfort evoked in this study should not go beyond mild levels of stress. If your stress or discomfort levels become uncomfortably high at any time during the study, please notify your experimenter at once and the study will stop immediately. If needed, the experimenter can refer you to a counselor.

I understand that each in-lab session will take 1.5 - 2 hours (on seven separate occasions: baseline assessment day 1 & 2, laptop instruction session, 1-month post assessment day 1 & 2, and 12-month follow-up assessment day 1 & 2). A full completion of this study will result in a payment rate of \$40 for completion of each assessment (the baseline / 1-month post / 12-month follow-up) and \$20 for the laptop instruction session for a total of \$140.

I understand that this study is registered in ClinicalTrials.gov (https://clinicaltrials.gov/). Running it as a clinical trial is intended to further protect the safety of the participants and ensure the quality and validity of research protocols. I also understand that according to Clinical Trials protocol, the study results and de-identified data (using participant numbers not names) will be reported to ClinicalTrials.gov.

I understand that this consent may be withdrawn at any time without prejudice, penalty or loss of benefits to which I am otherwise entitled. Partial completion will be compensated \$10 per hour. I have been given the right to ask and have answered any inquiry concerning the study. Questions, if any, have been answered to my satisfaction. I understand that I may decline to answer any question presented during this study.

I grant researchers the right to contact me for future related studies, and I have the right to accept or decline those requests. I understand that I may contact the project principal investigator, Dr. Walter Boot, Florida State University, Department of Psychology, 1107 W Call St., Tallahassee, Florida 32306-2540, (850) 644-6686, (boot@psy.fsu.edu) or Professor Neil Charness, (850) 644-6686 (charness@psy.fsu.edu) for answers to questions about this research. I understand I can also contact the Florida State University Office of Research, Human Subjects Committee, 2010 Levy Ave Research Building B Suite 276, Tallahassee, FL 32306, (850) 644-8673, (humansubjects@magnet.fsu.edu) with any grievances. The results of the study will be sent to me upon my request.

| l have read a<br>valid driver's | onsent form. I | am 18 years of age or older and ha | ve |
|---|---|---|---|
| Name | | Date | _ |

а

FSU Human Subjects Committee approved on 04/23/18. Void after 04/22/19. HSC # 2018.23703